CLINICAL TRIAL: NCT01955252
Title: Effect of WHO-yaws Elimination Strategy in Lihir Island, Papua New Guinea
Acronym: YESA-13
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lihir Medical Centre (Other)
Collaborators: Barcelona Institute for Global Health (Other); National Department of Health of Papua New Guinea (Unknown); World Health Organization (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Oriol Mitja, Community Health Director, Lihir Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YESA-13
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-01

CONDITIONS: Yaws
Keywords: Endemic treponematoses; Azithromycin; Mass drug administration; Eradication
MeSH Terms: conditions — Yaws | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azithromycin (Experimental): All participants older than 2 months (population 18,000) will be offered a single oral dose of oral azithromycin (tablets) 30 mg per Kg up to a maximum dose of 2g.
  Women who tell the investigators they are pregnant and people with known allergy to macrolides will be offered benzathine benzylpenicillin.
  This will be a single arm study. Study participants who met the inclusion criteria and agree to sign the consent form will be managed with proposed drug and systematically observed to measure outcomes of interest.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Investigators will do a baseline survey of every children from 5 to 15 years in the village. To detect yaws infection, investigators will collect a blood specimen for serology (qualitative and quantitative RPR testing and TPHA assay).
  Investigators will identify yaws-like ulcers by means of dermatological examination. Investigators will swab papilloma and ulcers and specimens will be flown to University of Washington (Seattle). PCR methods will consist of primary screening for the presence or absence of T. p. pertenue DNA, Haemophilus ducreyi DNA and detection of the A2058G and A2059G mutations associated with azithromycin resistance.
  Investigators will begin treatment with antibiotics immediately after completion of the baseline survey. Everyone in the villages will be offered azithromycin, subsequently a field team will treat all active clinical cases and their contacts 6 monthly.
  For all subjects, follow-up examination will be performed at 6,12,18,24,30,36,40,and 42 months
  Other Names: Azithromycin tablets 500mg (Medopharm); Zithromax

SUMMARY:
The trial that the investigators are proposing is a pilot study to determine the effect of the new WHO-yaws eradication strategy in Lihir Island (population 18,000), Papua New Guinea. New treatment policies were developed by WHO in 2012 to replace those of the 1950s. The recommended practice is to offer an initial MDA with azithromycin to the entire population, followed by resurveys every 6 months to detect and treat remaining cases.We will use serology surveys, clinical surveys and ulcer aetiology studies to measure the effect of mass azithromycin treatment on the community burden of yaws infection.

DETAILED DESCRIPTION:
Yaws is a re-emerging endemic treponemal infection caused by Treponema pallidum subp pertenue. This bacterium causes a chronic relapsing disease, characterized by highly contagious primary and secondary cutaneous lesions and non-contagious tertiary late destructive lesions. The Pacific Islands are believed to be a major focus of yaws worldwide, though population-based data on prevalence are lacking for many countries.

Azithromycin (30mg/kg) has recently been shown to be effective in the treatment of yaws and is now central to WHO's yaws eradication strategy. Substituting a single dose of an oral antibiotic for a painful penicillin injection is a significant advantage because infection control measures required for injection of penicillin will no longer be required and treatment will be more acceptable to communities who need it.

Previous attempts to eradicate yaws by mass treatment of active cases with injectable drugs yielded unsuccessful results. A major campaign to eradicate yaws in the 1950s and 1960s with longacting, injectable penicillin greatly reduced the number of cases of the disease worldwide but incubating and latent cases that were not treated developed relapses with infectious yaws lesions, thereby becoming a source of reinfection.

While the earlier strategy in the 1950s, targeted just those people who were visibly infected, the new WHO-plan calls for blanket coverage of at least 90% of the population. The ratio of clinically apparent to latent cases with no symptoms is estimated as high as 1:6 and mass drug administration (MDA) of the entire population is the best approach to ensure that incubating and latent infections are adequately dealt with.

The currently recommended treatment for eradication is one dose of oral azithromycin (30 mg/Kg; maximum 2g) to be given to entire populations in areas known to harbor yaws. For the MDA to be effective, it is required to have substantial coverage in the first round. The initial mass treatment should be followed by resurveys every 6 months to detect and treat remaining cases.

Because of the potential bacterial resistance appearance treatment failure needs to be monitored. Macrolide resistance is associated with point mutations at positions A2058 and A2059 of the 23S ribosomal RNA gene and molecular analysis need to be done in clinical specimens from patients who do not respond to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Whole resident population for MDA and clinical surveys, and children 5-15 years in sentinel sites for cross-sectional serological surveys.

Exclusion Criteria:

* Children younger than 2 months and pregnant women;
* Known allergy to macrolide antibiotics;
* Refusal of individual or guardian (for individual inclusion).

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16000 (Actual)
Dates: Start 2013-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of yaws latent infection | 42 months
  Prevalence of yaws infection is determined by the combination of a positive TPHA and RPR titer of 1:4 or above (which can be considered as the marker for true disease) in 1200 children 5-15 years in 6 randomly selected villages.

SECONDARY OUTCOMES:
Prevalence of active yaws disease | 42 months
  Determined by means of dermatological examination (WHO definitions) with laboratory confirmation using serology and PCR methods.
Macrolide resistance | 42 months
  Estimate the prevalence of molecular markers of macrolide resistance in T. pallidum subsp. pertenue in patients with active yaws both before and after the mass drug administration.
Ulcer aetiology surveys | 42 months
  PCR-surveillance of yaws-like ulcers in randomly selected villages every survey. This will allow to compare the relative proportion of T. pallidum pertenue ulcers vs other aetiological agents

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Mitja, MD, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (1):
- Lihir Medical Centre, Londolovit, New Ireland Province, Papua New Guinea

REFERENCES:
- [Derived] Mitja O, Godornes C, Houinei W, Kapa A, Paru R, Abel H, Gonzalez-Beiras C, Bieb SV, Wangi J, Barry AE, Sanz S, Bassat Q, Lukehart SA. Re-emergence of yaws after single mass azithromycin treatment followed by targeted treatment: a longitudinal study. Lancet. 2018 Apr 21;391(10130):1599-1607. doi: 10.1016/S0140-6736(18)30204-6. Epub 2018 Feb 7. PMID 29428183
- [Derived] Mitja O, Gonzalez-Beiras C, Godornes C, Kolmau R, Houinei W, Abel H, Kapa A, Paru R, Bieb SV, Wangi J, Sanz S, Asiedu K, Lukehart SA, Bassat Q. Effectiveness of single-dose azithromycin to treat latent yaws: a longitudinal comparative cohort study. Lancet Glob Health. 2017 Dec;5(12):e1268-e1274. doi: 10.1016/S2214-109X(17)30388-1. Epub 2017 Oct 26. PMID 29107621
- [Derived] Mitja O, Houinei W, Moses P, Kapa A, Paru R, Hays R, Lukehart S, Godornes C, Bieb SV, Grice T, Siba P, Mabey D, Sanz S, Alonso PL, Asiedu K, Bassat Q. Mass treatment with single-dose azithromycin for yaws. N Engl J Med. 2015 Feb 19;372(8):703-10. doi: 10.1056/NEJMoa1408586. PMID 25693010